CLINICAL TRIAL: NCT02702687
Title: Childhood Asthma Perception Study
Acronym: CAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-3257; 1R01HL128260-01 (NIH)
Record Dates: First submitted 2016-02-25; First posted 2016-03-09 (Estimated); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Asthma; Childhood Asthma
Keywords: Asthma; Childhood Asthma; Bronchial Diseases; Immune System Diseases; Lung Diseases; Lung Diseases, Obstructive; Respiratory Tract Diseases; Peak Flow Meter; Symptom Perception; Illness Representation
MeSH Terms: conditions — Asthma; Bronchial Diseases; Immune System Diseases; Lung Diseases; Lung Diseases, Obstructive; Respiratory Tract Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PEF Feedback (Experimental): This group will have 9 visits across 15 months.
  Interventions: Behavioral: PEF Feedback
- Control Feedback (Active Comparator): This group will have 9 visits across 15 months.
  Interventions: Behavioral: Control Feedback

INTERVENTIONS:
Behavioral: PEF Feedback — Intervention group will receive PEF feedback and verbal feedback sessions across 3 feedback visits and asthma education.
  Arms: PEF Feedback
Behavioral: Control Feedback — Control feedback group will receive feedback consisting of standardized messages and have 3 control feedback visits and asthma education.
  Arms: Control Feedback

SUMMARY:
This randomized controlled trial will include Latino and Black adolescents with asthma ages 10-17 years old and their caregivers. Participants will be recruited from clinics in the Bronx, New York. The primary aims are to examine the efficacy of peak expiratory flow (PEF) prediction with feedback versus control feedback on 1) under-perception of asthma symptoms 2) controller medication adherence and 3) asthma control and emergency health care use. These aims will be examined across a 1-year follow-up. An exploratory aim examines the hypothesized pathway that the PEF intervention reduces under-perception of symptoms, shifts illness representations toward the professional model and increases adolescents' and parents' asthma management self-efficacy, resulting in greater medication adherence and improved asthma control.

DETAILED DESCRIPTION:
Under-perception of asthma symptoms in children is a major risk factor for emergency department visits, hospitalizations, and near-fatal/fatal asthma attacks. Puerto Rican and Black children have greater asthma morbidity and mortality rates than all other racial/ethnic groups. Interventions targeting asthma symptom perception and medication adherence may help close this asthma health disparities gap.

The baseline visit for all families consists of standardized asthma education followed by 3 weeks of PEF prediction without feedback using a programmable, electronic spirometer. Participants then will be randomized to intervention group or control feedback group and receive a brief feedback session. For the next 6 weeks, all adolescents will predict their PEF, which will be locked in before blowing into the device. Families will return at mid-intervention and post-intervention to receive feedback sessions. All adolescents will play an interactive asthma educational game to reinforce the baseline asthma education. At the post-intervention visit, the spirometer will be reprogrammed for the next 4 weeks. These symptom perception data will be downloaded at 1-month post-intervention. Controller medication adherence will be monitored by electronic devices. Post-intervention sessions will take place at 3, 6, 9, and 12 months to collect adherence data and conduct spirometry. Physicians will be blinded to group assignment and rate asthma severity using national guidelines. A 12-month retrospective medical record abstraction will compare emergency health care use for asthma between groups.

ELIGIBILITY:
Inclusion Criteria:

* 10-17 years of age
* Diagnosis of asthma (in medical record)
* Report of breathing problems within the past 12 months
* Prescribed a controller medication for asthma
* At least one parent self-identifies as Latino or Black
* The participating parent has primary or at least equal responsibility for the adolescent

Exclusion Criteria:

* Cognitive learning disability (parent report)
* No prescription for asthma controller medication
* Inability to perform acceptable PEF blows
* Race/ethnicity other than Latino or Black
* Other significant pulmonary conditions (cystic fibrosis)

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 363 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
Asthma Symptom Perception with Asthma Monitor (AM2) as percentage of guesses in the Under-Perception zone | Change from Pre-intervention to 12-month-follow-up (15 months)
  The percentage of times a child under-perceives the severity of asthma symptoms

SECONDARY OUTCOMES:
Asthma Illness Representation Scale (AIRS) | Change from Pre-intervention to 12-month-follow-up (15 months)
  37-item scale measuring risk factors for the underutilization of controller medications
Asthma Management Self-Efficacy (ASE) scale: Parent and child versions | Change from Pre-intervention to 12-month-follow-up (15 months)
  13-item scale measures parent's confidence in their ability to help manage child's asthma
Pediatric Asthma Quality of Life Questionnaire (PAQLQ) | Change from Pre-intervention to 12-month-follow-up (15 months)
  23-item self report questionnaire assessing child's overall functioning in relation to asthma
Medication Adherence - percentage of total doses taken per day/prescribed per day | Change from Pre-intervention to 12-month-follow-up (15 months)
  Self report of daily medication use, in relation to the prescribed use
Health Care Use - Electronic Medical Record (EMR) review of asthma-related Emergency Department visits and hospitalizations | Change from Pre-intervention to 12-month-follow-up (15 months)
  Quantity of asthma-related emergency visits throughout the duration of the study
Asthma Control Test (C-ACT) | Change from Pre-intervention to 12-month-follow-up (15 months)
  Self-report questionnaire for adolescents and parents

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Feldman, PhD, Principal Investigator — Albert Einstein College of Medicine
Locations (2):
- United States (2):
  - Jacobi Medical Center, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feldman JM, Rastogi D, Warman K, Serebrisky D, Arcoleo K. Peak Flow Feedback Intervention Improves Underperception of Airflow Limitation in Pediatric Asthma: A Randomized Clinical Trial. Ann Am Thorac Soc. 2025 Mar;22(3):403-415. doi: 10.1513/AnnalsATS.202406-637OC. PMID 39454196

DOCUMENTS (1):
  • Informed Consent Form (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/87/NCT02702687/ICF_000.pdf